CLINICAL TRIAL: NCT07014709
Title: Impact of GLP-1 Receptor Agonists on Patients With Intraductal Papillary Mucinous Neoplasms: A Retrospective Multicentric Cohort Study
Brief Title: Impact of GLP-1 Receptor Agonists on Patients With IPMN
Acronym: IPMN-GLP1RA
Status: Not yet recruiting | Type: Observational
Sponsor: Hôpital Fribourgeois (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other); University Hospital, Geneva (Other)
Responsible Party: Sponsor
Other Study IDs: IPMN-GLP1RA
Record Dates: First submitted 2025-04-30; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: IPMN; IPMN, Pancreatic; GLP-1; Intraductal Papillary Mucinous Neoplasm of Pancreas; Glucagon-Like Peptide-1 Receptor Agonists
MeSH Terms: conditions — Pancreatic Intraductal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intraductal Papillary Mucinous Neoplasms: Patients eligible for this study must have a radiological diagnosis of IPMN
  Interventions: Drug: GLP1 receptor agonist

INTERVENTIONS:
Drug: GLP1 receptor agonist — Patients must be under GLP1-RA treatment for ether diabetes or obesity

SUMMARY:
This study investigates the impact of GLP-1 receptor agonists (GLP-1 RAs) on patients with intraductal papillary mucinous neoplasms (IPMNs), a type of pancreatic cystic neoplasm that can progress to malignancy. With the increasing use of GLP-1 RAs for managing diabetes and obesity, concerns about their potential to influence pancreatic conditions, like IPMNs, have emerged. Although GLP-1 RAs are generally safe, their effects on pre-existing pancreatic conditions remain unclear.

The study aims to evaluate whether GLP-1 RA use in IPMN patients is linked to changes in pancreatic cyst characteristics, the incidence of acute pancreatitis, variations in tumor markers, and the progression of IPMNs to high-grade dysplasia or malignancy. A retrospective analysis will be conducted using medical data from patients diagnosed with IPMNs and treated with GLP-1 RAs between 2010 and 2024 at three Swiss hospitals. Key outcomes will include radiological changes, the incidence of acute pancreatitis, and potential shifts in IPMN surveillance or need for surgical intervention

DETAILED DESCRIPTION:
This is a retrospective, multicentric cohort study designed to investigate the impact of GLP-1 receptor agonists (GLP-1 RAs) on patients with intraductal papillary mucinous neoplasms (IPMNs), a subtype of pancreatic cystic neoplasms with variable but potentially significant malignant potential. IPMNs are increasingly diagnosed due to advancements in cross-sectional imaging techniques, and their management often includes long-term radiological and clinical surveillance.

Concurrently, the prescription of GLP-1 RAs for type 2 diabetes mellitus and obesity has grown substantially. While GLP-1 RAs have shown excellent efficacy in glycemic control and weight reduction, concerns persist regarding their potential effects on the exocrine pancreas, particularly in patients with preexisting pancreatic abnormalities. Preclinical data in rodent models have been inconsistent, showing both pro-inflammatory and anti-inflammatory effects on the pancreas. Moreover, changes in pancreatic ductal morphology, including ductal gland proliferation, have been reported in animal studies, but with limited translation to human models. Meta-analyses of human clinical trials have not established a conclusive association between GLP-1 RAs and acute pancreatitis or pancreatic cancer; however, these studies typically exclude patients with underlying pancreatic lesions, such as IPMNs.

To address this gap, this study aims to assess the real-world effects of GLP-1 RA therapy on patients diagnosed with IPMNs. The hypothesis driving this research is that GLP-1 RA use may influence IPMN characteristics or related outcomes, which could affect management decisions including surveillance intervals, imaging modality choice, and surgical indications.

Study Setting and Data Sources The study is being conducted across 3 major Swiss medical centers: Hôpital Fribourgeois (HFR), Hôpitaux Universitaires de Genève (HUG), and the Inselspital in Bern. Data will be extracted from electronic medical records and include radiological images, laboratory test results, medication history, and clinical notes. The retrospective inclusion period ranges from January 2010 to May 2025.

Study Population Eligible participants are adult patients (aged ≥18 years) with a radiological diagnosis of IPMN who have been treated with any GLP-1 RA (e.g., exenatide, liraglutide, dulaglutide, semaglutide) during the study period. IPMN diagnoses will be validated based on radiologic criteria, with reference to the Kyoto 2023 Consensus. Patients must have complete medical records including at least one cross-sectional imaging (MRI or CT), serum tumor markers (CA19-9, CEA), and documented use of a GLP-1 RA.

Data Collection and Variables Collected variables include demographic information (age, sex, BMI), medical history (including diabetes subtype and comorbidities), GLP-1 RA treatment details (agent, dose, duration), laboratory values (HbA1c, fasting glucose, insulin, C-peptide, CA19-9, CEA, lipase, amylase), imaging features (cyst morphology, mural nodules, duct dilation), and clinical outcomes (acute pancreatitis, histopathologic progression, surveillance or surgical changes).

Radiological Evaluation All imaging studies will be re-reviewed by two independent, senior radiologists at HFR. Radiologists will be blinded to GLP-1 RA exposure. MRI is preferred; CT scans will be evaluated when MRI is unavailable. Radiological criteria from the Kyoto 2023 Consensus will be used, including assessment of cyst size, mural nodules, main duct diameter, enhancement features, and glandular morphology.

Statistical Analysis Descriptive statistics will be used to summarize baseline characteristics. Chi-square or Fisher's exact tests will be used for categorical variables, and t-tests or Mann-Whitney U tests for continuous variables. Multivariable logistic regression will control for potential confounders. Significance will be set at p < 0.05. A formal power calculation is not possible due to the exploratory and rare nature of the cohort, but the estimated sample size is 10-15 patients.

Data Quality and Management Data will be coded and entered into a centralized, secure RedCap database. Only authorized users will access the data. All changes will be tracked with an audit trail. Data validation procedures will include logic checks, range checks, and cross-field consistency. Periodic internal monitoring will be conducted to ensure protocol adherence.

Ethical Considerations All participating centers have received approval from their respective ethics committees. Patients provided general consent for use of anonymized medical data in research. Data will be anonymized and securely stored in compliance with Swiss data protection laws.

Expected Impact This study addresses an important clinical question that has not yet been explored in the literature. Its findings will help inform clinicians on whether GLP-1 RAs are safe for use in patients with IPMNs, potentially affecting surveillance strategies and therapeutic decisions. Results are expected to guide future prospective studies and could influence clinical guidelines related to pancreatic cystic lesions in patients with metabolic disease.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* Radiological diagnosis of IPMN
* Treated with GLP-1 RAs.
* Patients must have provided prior informed consent for the use of their coded clinical data in research.

Exclusion Criteria:

* radiological diagnosis of IPMN is unclear,
* no documented history of GLP-1 RAs use
* patients did not provide signed informed consent, or have documented refusal for research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients diagnosed with intraductal papillary mucinous neoplasms (IPMNs) who have been treated with GLP-1 receptor agonists (GLP-1 RAs) for diabetes or obesity management
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-05-31 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Radiological changes in pancreatic cyst characteristic as described in the Kyoto 2023 Consensus | during the GLP1 RA treatment
  Radiological data, including data from MRI scans, will be used to monitor changes in IPMN characteristics. If only CT scans are available, they will also be evaluated, even if this is not the preferred imaging method for IPMN evaluation

SECONDARY OUTCOMES:
Incidence of acute pancreatitis | during the GLP1 RA treatment
  The incidence of acute pancreatitis under GLP1-RA will be evaluated
Changes in serum tumor markers, CA19-9 and CEA levels | during the GLP1 RA treatment
  When already available in routine analyses before and after initiation of GLP-1 RA therapy, tumor markers level will be assessed to detect any changes
Changes in Endoscopic ultrasonography (EUS) characteristics | during the GLP1 RA treatment
  Evaluate the changes of morphological IPMN characteristic in endoscopic ultrasonography (EUS)
Progression of IPMNs to high-grade dysplasia or invasive malignancy in histopathological analysis | during the GLP1 RA treatment
  Evaluate the progression of IPMNs to high-grade dysplasia or invasive malignancy in histopathological analysis
Need for surgical intervention | during the GLP1 RA treatment
  Investigate the need for surgical intervention associated with the introduction of GLP-1 RA treatment
Changes in IPMN surveillance protocols | during the GLP1 RA treatment
  Investigate the need for changes in IPMN surveillance protocols associated with GLP-1 RA use.

CONTACTS AND LOCATIONS:
Locations (1):
- HFR Hopital fribourgeois, Villars-sur-Glâne, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ohtsuka T, Fernandez-Del Castillo C, Furukawa T, Hijioka S, Jang JY, Lennon AM, Miyasaka Y, Ohno E, Salvia R, Wolfgang CL, Wood LD. International evidence-based Kyoto guidelines for the management of intraductal papillary mucinous neoplasm of the pancreas. Pancreatology. 2024 Mar;24(2):255-270. doi: 10.1016/j.pan.2023.12.009. Epub 2023 Dec 28. PMID 38182527